CLINICAL TRIAL: NCT00052221
Title: A Placebo Controlled Trial Of Short-Term, High-Dose Epoetin Alfa In Advanced Cancer Outpatients With Mild Fatigue
Brief Title: Epoetin Alfa in Treating Fatigue in Patients With Advanced Solid Tumors Who Are Not Receiving Chemotherapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CDR0000069409; MDA-DM-02331; MDA-DM-0038; NCI-P02-0225; DM02-331 (Other: UT MD Anderson Cancer Center); NCT00563719 (obsolete NCT alias)
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Fatigue; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; fatigue
MeSH Terms: conditions — Fatigue | interventions — Epoetin Alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I: Epoetin Alfa (Experimental): Epoetin alfa subcutaneously (SC) once weekly for 6 weeks
  Interventions: Biological: Epoetin alfa
- Arm II: Placebo (Placebo Comparator): Placebo subcutaneously (SC) once weekly for 6 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Epoetin alfa
  Arms: Arm I: Epoetin Alfa
Other: Placebo
  Arms: Arm II: Placebo

SUMMARY:
RATIONALE: Epoetin alfa may help improve energy levels and quality of life in patients who have advanced solid tumors.

PURPOSE: Randomized clinical trial to study the effectiveness of epoetin alfa in treating fatigue in patients who are not receiving chemotherapy for advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of epoetin alfa in treating fatigue in patients with advanced solid tumors who are not receiving chemotherapy.
* Determine the efficacy of this drug on functional status and overall quality of life in these patients.
* Correlate self-reported level of energy with other commonly occurring symptoms (e.g., pain, depression, anxiety, dyspnea, appetite disturbance, or sleep disturbance) in these patients.
* Correlate anemia with other common symptoms in these patients.
* Determine the internal consistency of fatigue self-report using three single-item measures of this symptom and the responsiveness of each item to change over time in these patients.

OUTLINE: This is a double-blind, placebo-controlled, randomized, multicenter study. Patients are stratified according to participating center, ECOG performance status (0-1 vs 2-3), and hemoglobin prior to study (10 mg/dL or less vs greater than10 mg/dL). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive epoetin alfa subcutaneously (SC) once weekly for 6 weeks.
* Arm II: Patients receive placebo SC once weekly for 6 weeks. Patients in either arm that do not respond to therapy may receive an additional 6 weeks of open-label epoetin alfa SC once weekly.

In both arms, quality of life and fatigue are assessed at baseline and at 3 and 6 weeks. If patients receive an additional 6 weeks of therapy, quality of life and fatigue are also assessed at 9 and 12 weeks.

PROJECTED ACCRUAL: A total of 128 patients (64 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of stage III or IV invasive non-myeloid malignancy
* Not currently hospitalized
* At least somewhat bothered by fatigue based on self-report

  * No significant psychological distress indicated by total score of 6 or more on questions 1 and 2 of the Three-Question Screening Survey (3QSS)
  * No score less than 2 on question 3 of 3QSS indicating low level of fatigue within the past week
* No uncontrolled brain metastases or leptomeningeal involvement

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Eastern Cooperative Oncology Group (ECOG) 0-3

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Hemoglobin at least 8.5 g/dL but no greater than 11 g/dL
* No anemia due to factors other than cancer or chemotherapy (e.g., iron or folate deficiency, hemolysis, or bleeding)
* No prior or concurrent hematological disease

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* No uncontrolled hypertension (diastolic blood pressure greater than 100 mm Hg or systolic blood pressure greater than 200 mm Hg)
* No significant uncontrolled concurrent cardiovascular disease or dysfunction not attributable to malignancy or chemotherapy
* No history of deep-vein thrombosis

Pulmonary:

* No significant uncontrolled concurrent pulmonary disease or dysfunction not attributable to malignancy or chemotherapy

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 3 months after study participation
* Able to understand and complete self-report symptom assessment forms in English
* No serious concurrent infection
* No known hypersensitivity to mammalian cell-derived products or human albumin
* No uncontrolled seizures
* No significant uncontrolled concurrent endocrine, neurologic, gastrointestinal, or genitourinary system disease or dysfunction not attributable to malignancy or chemotherapy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Chemotherapy
* More than 4 weeks since prior biologic therapy (e.g., interferon or interleukin-2)
* More than 2 months since prior red blood cells (RBC) transfusion
* More than 1 month since prior epoetin alfa or investigational forms of epoetin alfa (e.g., gene-activated, novel erythropoiesis-stimulating protein)
* Concurrent non-myelosuppressive therapy (e.g., monoclonal antibody infusions, antiangiogenesis inhibitors, or signal transduction inhibitors) allowed
* No other concurrent biologic therapy

Chemotherapy:

* No prior high-dose chemotherapy (e.g., with bone marrow or stem cell transplantation)
* More than 4 weeks since prior chemotherapy
* No concurrent chemotherapy

Endocrine therapy:

* Concurrent hormonal therapy allowed (e.g., luteinizing hormone-releasing hormone agonists or tamoxifen)

Radiotherapy:

* More than 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2003-05-20 (Actual); Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Fisch, MD, MPH, FACP, Study Chair — M.D. Anderson Cancer Center